CLINICAL TRIAL: NCT00025337
Title: Phase III Trial of Bevacizumab (NSC 704865), Oxaliplatin (NSC 266046), Fluorouracil and Leucovorin Versus Oxaliplatin, Fluorouracil and Leucovorin Versus Bevacizumab Alone in Previously Treated Patients With Advanced Colorectal Cancer
Brief Title: Combination Chemotherapy With or Without Bevacizumab Compared With Bevacizumab Alone in Treating Patients With Advanced or Metastatic Colorectal Cancer That Has Been Previously Treated
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02417; E3200; U10CA021115 (NIH); CDR0000068951 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage III Colon Cancer; Stage III Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Leucovorin; Fluorouracil

ARMS (3):
- Arm I (bevacizumab, oxaliplatin, leucovorin, fluorouracil) (Experimental): Patients receive bevacizumab IV over 30-90 minutes and oxaliplatin IV over 2 hours on day 1. Patients also receive leucovorin calcium IV over 2 hours and fluorouracil (5-FU) IV over 22 hours on days 1 and 2.
  Interventions: Biological: bevacizumab; Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil
- Arm II (oxaliplatin, leucovorin calcium, fluorouracil) (Experimental): Patients receive oxaliplatin, leucovorin calcium, and 5-FU as in arm I.
  Interventions: Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil
- Arm III (bevacizumab) (Experimental): Patients receive bevacizumab as in arm I.
  Interventions: Biological: bevacizumab

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
  Arms: Arm I (bevacizumab, oxaliplatin, leucovorin, fluorouracil); Arm III (bevacizumab)
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
  Arms: Arm I (bevacizumab, oxaliplatin, leucovorin, fluorouracil); Arm II (oxaliplatin, leucovorin calcium, fluorouracil)
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
  Arms: Arm I (bevacizumab, oxaliplatin, leucovorin, fluorouracil); Arm II (oxaliplatin, leucovorin calcium, fluorouracil)
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
  Arms: Arm I (bevacizumab, oxaliplatin, leucovorin, fluorouracil); Arm II (oxaliplatin, leucovorin calcium, fluorouracil)

SUMMARY:
Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without bevacizumab in treating patients who have advanced or metastatic colorectal cancer that has been previously treated. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as bevacizumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining monoclonal antibody therapy with combination chemotherapy may kill more tumor cells. It is not yet known if bevacizumab is more effective with or without combination chemotherapy in treating colorectal cancer

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the response, time to progression, and overall survival of patients with previously treated advanced or metastatic colorectal adenocarcinoma treated with oxaliplatin, leucovorin calcium, and fluorouracil with or without bevacizumab versus bevacizumab only. (Arm III closed to accrual as of 03/11/2003).

II. Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to ECOG performance status (0 vs 1 or 2), and prior radiotherapy (yes vs no). Patients are randomized to 1 of 3 treatment arms.

Arm I: Patients receive bevacizumab IV over 30-90 minutes and oxaliplatin IV over 2 hours on day 1. Patients also receive leucovorin calcium IV over 2 hours and fluorouracil (5-FU) IV over 22 hours on days 1 and 2.

Arm II: Patients receive oxaliplatin, leucovorin calcium, and 5-FU as in arm I.

Arm III: Patients receive bevacizumab as in arm I. (Arm closed to accrual as of 03/11/2003).

Courses in all arms repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response may receive 2 additional courses.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the colon or rectum

  * Advanced or metastatic disease
  * Must have received a fluoropyrimidine-based regimen and an irinotecan-based regimen, either alone or in combination, for advanced disease
  * May have relapsed within 6 months of adjuvant therapy with fluorouracil (5-FU) (or combination 5-FU and irinotecan) and progressed after single-agent irinotecan
* Measurable disease
* No known brain metastases
* Performance status - ECOG 0-2
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No history of thrombotic or hemorrhagic disorders
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 5 times ULN
* INR no greater than 1.5
* PTT no greater than ULN
* Creatinine no greater than 1.5 times ULN
* Proteinuria less than 1+ (i.e., 0 or trace)
* Protein less than 500 mg by 24-hour urine collection
* Proteinuria secondary to ureteral stents allowed

  * No proteinuria secondary to nephropathy
* Controlled hypertension (less than 150/100 mm Hg) allowed if on a stable antihypertensive regimen
* No prior myocardial infarction
* No uncontrolled congestive heart failure
* No unstable angina within the past 3 months
* No serious nonhealing wound, ulcer, or bone fracture
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior bevacizumab
* See Disease Characteristics
* Recovered from prior chemotherapy
* No prior oxaliplatin
* At least 2 weeks since prior radiotherapy and recovered
* At least 28 days since prior major surgical procedure
* At least 10 days since prior aspirin dose of more than 325 mg/day
* No concurrent therapeutic anticoagulation except prophylactic anticoagulation of venous access device
* No concurrent antiplatelet agents (e.g., dipyridamole, ticlopidine, clopidogrel, or cilostazol)
* No concurrent oral cryotherapy on day 1 of oxaliplatin administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Actual)
Dates: Start 2001-09; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Overall survival | From the date of entry on study, assessed up to 5 years

SECONDARY OUTCOMES:
Response defined using RECIST criteria | Up to 5 years
Progression free survival | From the date of entry on the study to the appearance of new metastatic lesions or objective tumor progression, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Giantonio, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States